CLINICAL TRIAL: NCT02297204
Title: Long-Term Efficacy and Safety of Intravitreal Aflibercept Injections for the Treatment of Diabetic Macular Edema in Subjects Who Completed the Three Year VISTA-DME Trial (The Endurance 1 Trial)
Brief Title: The Endurance 1 Trial
Acronym: Endurance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern California Retina Vitreous Associates (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Rahul Khurana, M.D., Principal Investigator, Northern California Retina Vitreous Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REG-2014-11-006; NCT02368756 (obsolete NCT alias)
Record Dates: First submitted 2014-11-14; First posted 2014-11-21 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aflibercept (Experimental): 2mg, as needed, intravitreal administration. All subjects will be treated with intravitreal (IVT) aflibercept injections as needed in the presence of clinically relevant diabetic macular edema (CR-DME). If CR-DME is not present the subject will not receive an IVT aflibercept injection and will be observed.
  If a subject has recurrent CR-DME they will receive an IVT aflibercept 2.0 mg injection and interval between visits will be reduced to 4 weeks.
  At week 12 through end of study, all subjects will be evaluated for focal laser treatment.
  Interventions: Procedure: Focal Laser Treatment; Drug: aflibercept 2.0 mg

INTERVENTIONS:
Procedure: Focal Laser Treatment — All subjects receiving PRN IVT aflibercept injections will be evaluated for focal laser treatment beginning at week 12 through the end of the study. If the subject meets any of the criteria for focal laser treatment (FLT), fluorescein angiography (FA) will be performed to guide the focal laser treatment. Focal laser treatment and focal laser re-treatment will be administered no more than once every 90 days.
  Other Names: FLT
Drug: aflibercept 2.0 mg — If a subject has recurrent CR-DME they will receive an IVT aflibercept injection
  Other Names: Eylea

SUMMARY:
The Endurance Trial is a phase IV open label clinical study to assess the need for ongoing intravitreal aflibercept injections after the 3-year VISTA DME (VGFT-OD-1009) end-point. Subjects will be treated with intravitreal aflibercept injections pro re nata (PRN) based on the presence of CR-DME (Clinically Relevant-Diabetic Macular Edema). In addition, subjects who meet re-treatment criteria will be eligible for focal laser treatment every 90 days.

DETAILED DESCRIPTION:
The safety and tolerability of intravitreal aflibercept injections have been investigated in previous Phase I, I/II and III studies in AMD, RVO, and DME trials. Potential safety issues associated with the route of administration or the pharmacology of aflibercept in the study population include decreased BCVA, intraocular inflammation, intraocular infection, transient and/or sustained elevation of intraocular pressure (IOP), cataract development or progression, retinal or intravitreal hemorrhage, macular edema, retinal break or detachment, and arterial thromboembolic events (ATEs). Safety will be assessed by visual acuity, ophthalmic examinations, fluorescein angiograms, OCT, intraocular pressure, vital signs, and adverse event documentation.

To minimize the risks of intraocular infections, all injections will be performed employing sterile techniques as described in Appendix A. Study drug administration will be held for subjects who experience certain ocular events or infections. In the event any subject develops an adverse event in the study eye that is considered by the evaluating physician to be severe in intensity, serious consideration should be given to withdrawing the subject from the study.

The PI or designated Sub-Investigators will review all adverse events on an ongoing basis to determine causality and relationship to study drug and/or study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled and Completed VISTA DME (VGFT-OD-1009) clinical trial
2. Willing and able to comply with clinic visits and study-related procedures
3. Provide signed informed consent
4. Enrollment in the trial within 12 weeks of trial activation.

Exclusion Criteria:

1. Prior treatment with anti-VEGF therapy in the study eye within 28 days of baseline
2. Pregnant or breast-feeding women
3. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly).

   * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11; Primary Completion 2017-12-13 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Need for ongoing intravitreal aflibercept injections in the management of DME | 12 months
  To assess the need for ongoing intravitreal aflibercept injections for subjects who were enrolled and completed the 3-year VISTA DME (VGFT-OD-1009) trial and to characterize long-term efficacy and safety of aflibercept intravitreal injections in the management of DME by evaluating mean number of injections in 52 weeks and proportion of subjects receiving 0 (zero) injections in 52 weeks.

SECONDARY OUTCOMES:
Vision change | 12 months
  Mean change in visual acuity from baseline to week 52.
Vision loss | 12 months
  Proportion of subjects with gain or loss of 0 to 5 letters from baseline to week 52.
Change in central retinal thickness | 12 months
  Mean change in central retinal thickness from baseline to week 52.
Development of clinically relevant diabetic macular edema | 12 months
  Percentage of subjects with no clinically relevant diabetic macular edema seen on SD-OCT from baseline to week 52
Role of focal laser treatment in management of DME (Proportion of subjects that receive focal laser treatment and mean number of intravitreal aflibercept injections before and after receiving focal laser treatment.) | 12 months
  Proportion of subjects that receive focal laser treatment and mean number of intravitreal aflibercept injections before and after receiving focal laser treatment.
Evaluation of Diabetic Retinopathy (Proportion of subjects with stable, worsened, or improved diabetic retinopathy as identified by eye examination and imaging.) | 12 months
  Proportion of subjects with stable, worsened, or improved diabetic retinopathy as identified by eye examination and imaging.
Ocular and systemic adverse events | 12 months
  Incidence and severity of ocular and systemic adverse events as identified by eye examinations, imaging, and subject reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Khurana, MD, Principal Investigator — Northern California Retina Vitreous Associates